CLINICAL TRIAL: NCT00997477
Title: A Single Arm, 12 Week, Multicentre, Open Label, Phase IV Study to Evaluate Correct Use of and Patient Satisfaction From Sequential Use of Formoterol and Budesonide Inhaler Capsules Via Aerolizer™ Device in Patients With Asthma.
Brief Title: Correct Use of Sequential Formoterol and Budesonide Inhaler Capsule Treatment Via Aerolizer and Patient Satisfaction in Asthmatics
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Medical Department, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFOR258FTR03
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2016-03

CONDITIONS: Asthma
Keywords: aerolizer; formoterol; budesonide; asthma
MeSH Terms: conditions — Asthma

ARMS (1):
- Formoterol and Budesonide (Experimental)
  Interventions: Drug: Foradil Combi (Formoterol-budesonide)

INTERVENTIONS:
Drug: Foradil Combi (Formoterol-budesonide)

SUMMARY:
This study will evaluate the correct use of sequential formoterol and budesonide inhaler capsule treatment via Aerolizer and patient satisfaction in adult asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* Moderate persistent asthmatic patients.
* No previous Aerolizer experience.

Exclusion Criteria:

* Life-threatening asthma: A subject must not have life-threatening asthma as a history of significant asthma episode(s)requiring intubation associated with hypercapnia, respiratory arrest or hypoxic seizures, or asthma-related syncopal episode(s).
* Worsening of asthma: A subject must not have experienced a worsening of asthma which involved a hospitalization within 6 months of screening, or an emergency room visit three or more times in the past 6 months, or use of oral corticosteroids for worsening asthma within 3 months of screening.
* Unstable asthma: During screening period, a patient requires the use of >8 puffs/day of salbutamol 100 mcg per actuation pMDI on two consecutive days.
* A subject must not have had an upper respiratory tract infection within 4 weeks of screening.
* FEV1< 60% at screening.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Proper use of Foradil Combi | Day 0, Day 30, Day 90

SECONDARY OUTCOMES:
Asthma control test | Day 0, Day 30, Day 90
Ease of use: FSI-10 Questionnaire | Day 30, Day 90
Patient Satisfaction: PSAM and FSI-10 | Evaluations will be made at visit 2 (Day 30± 1) and 3 (Day 90± 3)
Safety: Adverse events and severe adverse events | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Turkey (Türkiye) (4):
  - Novartis Investigator Site, Ankara
  - Novarits Investigator Site, Istanbul
  - Novartis Investigator Site, Istanbul
  - Novartis Investigator Site, Izmir